CLINICAL TRIAL: NCT02381496
Title: A Three-part Study to Assess the Tolerability, Safety, Pharmacodynamics, and Pharmacokinetics of Ascending Single Doses (Including Food Interaction) of ACT-453859 in Healthy Male Subjects, of Ascending Multiple Doses of ACT-453859 in Healthy Male and Female Subjects, and of Multiple Doses of Setipiprant (ACT-129968) in Healthy Male and Female Subjects
Brief Title: A Study to Assess the Tolerability, Safety, Pharmacodynamics, and Pharmacokinetics of Ascending Single Doses (Including Food Interaction) and Ascending Multiple Doses of ACT-453859, and Multiple Doses of Setipiprant (ACT-129968)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AC-072-101
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: ACT-453859; ACT-463036; Setipiprant; Tolerability; safety; pharmacodynamics; pharmacokinetics
MeSH Terms: interventions — ACT-453859; 2-(2-(1-naphthoyl)-8-fluoro-3,4-dihydro-1H-pyrido(4,3-b)indol-5(2H)-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- Part A: Cohort A1: ACT-453859 1 mg (Experimental): ACT-453859 1 mg or placebo, single dose, administered orally in the fasted state
  * Six male subjects will receive ACT-453859
  * Two male subjects will receive matching placebo
  Interventions: Drug: ACT-453859 1 mg; Other: Placebo
- Part A: Cohort A2: ACT-453859 3 mg (Experimental): ACT-453859 3 mg or placebo, single dose, administered orally in the fasted state
  * Six male subjects will receive ACT-453859
  * Two male subjects will receive matching placebo
  Interventions: Drug: ACT-453859 3 mg; Other: Placebo
- Part A: Cohort A3: ACT-453859 10 mg (Experimental): ACT-453859 10 mg or placebo, single dose, administered orally in the fasted state
  * Six male subjects will receive ACT-453859
  * Two male subjects will receive matching placebo
  Interventions: Drug: ACT-453859 10 mg; Other: Placebo
- Part A: Cohort A4: ACT-453859 30 mg (Experimental): ACT-453859 30 mg or placebo, single dose, administered orally in the fasted state
  * Six male subjects will receive ACT-453859
  * Two male subjects will receive matching placebo
  Interventions: Drug: ACT-453859 30mg; Other: Placebo
- Part A: Cohort A5: ACT-453859 100 mg (Experimental): ACT-453859 100 mg or placebo, single dose, administered orally in the fasted state
  * Six male subjects will receive ACT-453859
  * Two male subjects will receive matching placebo
  After a washout period of 10-20 days subjects will return for a second study period to receive the same treatment received in the first session but under fed conditions
  Interventions: Drug: ACT-453859 100 mg; Other: Placebo
- Part A: Cohort A6: ACT-453859 300 mg (Experimental): ACT-453859 300 mg or placebo, single dose, administered orally in the fasted state
  * Six male subjects will receive ACT-453859
  * Two male subjects will receive matching placebo
  Interventions: Drug: ACT-453859 300 mg; Other: Placebo
- Part A: Cohort A7: ACT-453859 800 mg (Experimental): ACT-453859 800 mg or placebo, single dose, administered orally in the fasted state
  * Six male subjects will receive ACT-453859
  * Two male subjects will receive matching placebo
  Interventions: Drug: ACT-453859 800 mg; Other: Placebo
- Part B: Cohort B1: ACT-453859 10 mg (Experimental): ACT-453859 10 mg or placebo, once a day for 7 days, administered orally in the fasted state
  * Three male subjects will receive ACT-453859
  * Three female subjects will receive ACT-453859
  * One male subject will receive matching placebo
  * One female subject will receive matching placebo
  Interventions: Drug: ACT-453859 10 mg; Other: Placebo
- Part B: Cohort B2: ACT-453859 100 mg (Experimental): ACT-453859 100 mg or placebo, once a day for 7 days, administered orally in the fasted state
  * Three male subjects will receive ACT-453859
  * Three female subjects will receive ACT-453859
  * One male subject will receive matching placebo
  * One female subject will receive matching placebo
  Interventions: Drug: ACT-453859 100 mg; Other: Placebo
- Part B: Cohort B3: ACT-453859 800 mg (Experimental): ACT-453859 800 mg, once a day for 7 days, administered orally in the fasted state
  * Three male subjects will receive ACT-453859
  * Three female subjects will receive ACT-453859
  * One male subject will receive matching placebo
  * One female subject will receive matching placebo
  Interventions: Drug: ACT-453859 800 mg; Other: Placebo
- Part C: Treatment Periods I & II: Setipiprant (Experimental): Setipiprant 500 mg, twice daily for 7 days, administered orally in Treatment Period I (TPI) and setipiprant 1000 mg, twice daily for 7 days, administered orally in Treatment Period II (TPII)
  * Four male subjects will receive setipiprant 500 mg twice a day in TPI and 1000 mg twice a day in TPII.
  * Four female subjects will receive setipiprant 500 mg twice a day in TPI and 1000 mg twice a day in TPII.
  There will be a washout period of 10 days between TPI and TPII
  Interventions: Drug: Setipiprant 500 mg; Drug: Setipiprant 1000 mg

INTERVENTIONS:
Drug: ACT-453859 1 mg — Capsule
  Arms: Part A: Cohort A1: ACT-453859 1 mg
Drug: ACT-453859 3 mg — Capsule
  Arms: Part A: Cohort A2: ACT-453859 3 mg
Drug: ACT-453859 10 mg — Capsule
  Arms: Part A: Cohort A3: ACT-453859 10 mg; Part B: Cohort B1: ACT-453859 10 mg
Drug: ACT-453859 30mg — Capsule
  Arms: Part A: Cohort A4: ACT-453859 30 mg
Drug: ACT-453859 100 mg — Capsule
  Arms: Part A: Cohort A5: ACT-453859 100 mg; Part B: Cohort B2: ACT-453859 100 mg
Drug: ACT-453859 300 mg — Capsule
  Arms: Part A: Cohort A6: ACT-453859 300 mg
Drug: ACT-453859 800 mg — Capsule
  Arms: Part A: Cohort A7: ACT-453859 800 mg; Part B: Cohort B3: ACT-453859 800 mg
Other: Placebo — Matching ACT-453859 placebo capsule
  Arms: Part A: Cohort A1: ACT-453859 1 mg; Part A: Cohort A2: ACT-453859 3 mg; Part A: Cohort A3: ACT-453859 10 mg; Part A: Cohort A4: ACT-453859 30 mg; Part A: Cohort A5: ACT-453859 100 mg; Part A: Cohort A6: ACT-453859 300 mg; Part A: Cohort A7: ACT-453859 800 mg; Part B: Cohort B1: ACT-453859 10 mg; Part B: Cohort B2: ACT-453859 100 mg; Part B: Cohort B3: ACT-453859 800 mg
Drug: Setipiprant 500 mg — Capsule
  Arms: Part C: Treatment Periods I & II: Setipiprant
Drug: Setipiprant 1000 mg — Capsule
  Arms: Part C: Treatment Periods I & II: Setipiprant

SUMMARY:
This is a three-part study to assess the tolerability, safety, pharmacodynamics, and pharmacokinetics of ascending single doses (including food interaction) of ACT-453859 in healthy male subjects, of ascending multiple doses of ACT-453859 in healthy male and female subjects, and of multiple doses of setipiprant (ACT-129968) in healthy male and female subjects.

DETAILED DESCRIPTION:
Part A of this study is a single-center, randomized, double-blind, placebo-controlled, single-ascending dose (SAD) design in healthy male subjects. In each cohort, eight subjects will be randomized as follows:

* Six male subjects will receive a single oral dose of ACT-453859, under fasted conditions.
* Two male subjects will receive matching placebo, under fasted conditions.

The doses of ACT-453859 were 1, 3, 10, 30, 100, 300, and 800 mg. Subjects in only one cohort (100 mg dose cohort) will come back for a second period of treatment under fed conditions.

Part B is a single-center, randomized, double-blind, placebo-controlled multiple-ascending dose (MAD) design in healthy male and female of subjects.

In each of 3 cohorts, eight subjects will be randomized to receive multiple doses of ACT-453859 or placebo once a day for 7 days as follows:

* Three male subjects will receive ACT-453859.
* Three female subjects will receive ACT-453859.
* One male subject will receive matching placebo.
* One female subject will receive matching placebo.

The doses of ACT-453859 will be 10, 100, and 800 mg per day.

Part C is a single-center and open-label design consisting of multiple oral doses of setipiprant given in a sequential design in healthy male and female subjects.

Eight subjects will be randomized to receive multiple doses of setipiprant for 7 days (only a single dose on Day 7), in Treatment Period I (TPI) and Treatment Period II (TPII), as follows:

* Four male subjects will receive setipiprant 500 mg twice a day (b.i.d.) in TPI and 1000 mg b.i.d. in TPII.
* Four female subjects will receive setipiprant 500 mg b.i.d. in TPI and 1000 mg b.i.d. in TPII.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Healthy male subjects (Part A), healthy male and female subjects for Parts B & C.
* Hematology, coagulation (Part A and Part B only), clinical chemistry, and urinalysis test results not deviating from the normal range to a clinically relevant extent.
* No clinically significant findings on physical examination.
* Body mass index between 18.0 and 28.0 kg/m^2.
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and heart rate 45-90 beats per minute.
* 12-lead electrocardiogram without clinically relevant abnormalities.
* Negative results from urine drug screen and alcohol breath test.
* Able and willing to refrain from sunbathing, prolonged sun exposure, and artificial sunlight exposure such as solarium, and to limit skin and eye exposure to sunlight using appropriate precautions from the first dose until safety follow-up visit for Parts A and B.
* Ability to communicate well with the investigator in the local language, and to understand and comply with the requirements of the study.
* For male subjects: consent that the female partner uses a medically acceptable method of contraception throughout the entire study period and for 90 days after the study is completed.
* For male subjects: agree not to donate sperm from the first drug administration until 90 days after completion of the study.
* For Part C, women of childbearing potential must have a negative serum pregnancy test and a negative urine pregnancy test pre-dose on Day 1 (of each treatment period for Part C). Women of childbearing potential must consistently and correctly use a reliable method of contraception, be sexually inactive or have a vasectomized partner.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Previous history of fainting, collapses, syncope, orthostatic hypotension, or vasovagal reactions.
* Veins unsuitable for intravenous puncture on either arm.
* Treatment with any prescribed or over-the-counter medications within 2 weeks prior to first study drug administration.
* Treatment or substances known to inhibit cytochrome P (CYP) enzyme drug metabolism .
* Treatment or substances known to induce CYP enzyme drug metabolism.
* Treatment with another investigational drug within 3 months prior or participated in more than four investigational drug studies within 1 year prior to Screening. Subjects will not participate in more than one part of the study.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to Screening.
* History or clinical evidence of any disease, and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs.
* Excessive caffeine consumption.
* Smoking, tobacco use, or use of nicotine products within 3 months and inability to refrain from smoking during the course of the study.
* Loss of 250 mL or more of blood, or an equivalent amount of plasma, within 3 months prior to Screening.
* Positive results from the hepatitis serology, except for vaccinated subjects or subjects with past but resolved hepatitis.
* Positive results from human immunodeficiency virus serology.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity.
* Pregnant or lactating women.
* Known allergic reactions or hypersensitivity to any excipients of the drug formulations.
* Difficulty in fasting or consuming standardized meals.
* Difficulty in swallowing whole tablets or capsules.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC(0-t)) for single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. AUC(0-t) will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification (LOQ).
AUC(0-t) for the active metabolite ACT-463036 after single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. AUC(0-t) will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the LOQ.
Area under the plasma concentration-time curve (AUC(0-infinity)) for single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. AUC(0-infinity) will be calculated by combining AUC(0-t) and AUC(extra). AUC(extra) represents an extrapolated value obtained by Ct/λz, where Ct is the last plasma concentration measured above the LOQ and λZ represents the terminal elimination rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal elimination phase.
AUC(0-infinity) for the active metabolite ACT-463036 after single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. AUC(0-infinity) will be calculated by combining AUC(0-t) and AUC(extra). AUC(extra) represents an extrapolated value obtained by Ct/λz, where Ct is the last plasma concentration measured above the LOQ and λZ represents the terminal elimination rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal elimination phase.
Time to reach maximum plasma concentration (tmax) for single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. The measured individual plasma concentrations of ACT-453859 will be used to directly obtain tmax.
tmax for the active metabolite ACT-463036 after single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. The measured individual plasma concentrations of ACT-463036 will be used to directly obtain tmax.
Terminal elimination rate constant (λZ) for single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. λZ will be determined by log-linear regression analysis of the measured plasma concentrations of the terminal elimination phase.
λZ for the active metabolite ACT-463036 after single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. λZ will be determined by log-linear regression analysis of the measured plasma concentrations of the terminal elimination phase.
Plasma half life (t1/2) for single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. t1/2 will be calculated as follows: t½ = ln 2/λZ.
t1/2 for the active metabolite ACT-463036 after single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. t1/2 will be calculated as follows: t½ = ln 2/λZ.
Maximum plasma concentration (Cmax) for single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. The measured individual plasma concentrations of ACT-453859 will be used to directly obtain Cmax.
Cmax for the active metabolite ACT-463036 after single doses of ACT-453859 | 72 hours
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. The measured individual plasma concentrations of ACT-463036 will be used to directly obtain Cmax.
Renal clearance (CLR) following single dose of ACT-453859 100 mg | 72 hours
  Urine samples for pharmacokinetic assessments will be collected at various time points over the study period. CLR will be calculated by dividing the total amount of unchanged ACT-453859 excreted in urine during the collection interval by AUC(0-t).
Percentage of ACT-453859 excreted unchanged in the urine following single dose of ACT-453859 100 mg | 72 hours
  Urine samples for pharmacokinetic assessments will be collected at various time points over the study period.The percentage of total dose excreted unchanged in urine will be calculated by the total amount excreted, divided by the dose administered, multiplied by 100.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUCτ) for multiple doses of ACT-453859 (Day 1 & Day 7) | 11 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. AUCτ will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the LOQ during one dosing interval.
AUCτ for the active metabolite ACT-463036 after multiple doses of ACT-453859 (Day 1 & Day 7) | 11 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. AUCτ will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the LOQ during one dosing interval.
Cmax for multiple doses of ACT-453859 (Day 1 & Day 7) | 11 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. The measured individual plasma concentrations of ACT-453859 will be used to directly obtain Cmax.
Cmax for the active metabolite ACT-463036 after multiple doses of ACT-453859 (Day 1 & Day 7) | 11 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. The measured individual plasma concentrations of ACT-463036 will be used to directly obtain Cmax.
tmax for multiple doses of ACT-453859 (Day 1 & Day 7) | 11 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. The measured individual plasma concentrations of ACT-453859 will be used to directly obtain tmax.
tmax for the active metabolite ACT-463036 after multiple doses of ACT-453859 (Day 1 & Day 7) | 11 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. The measured individual plasma concentrations of ACT-463036 will be used to directly obtain tmax.
λZ for multiple doses of ACT-453859 | 11 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. λZ will be determined by log-linear regression analysis of the measured plasma concentrations of the terminal elimination phase.
λZ for the active metabolite ACT-463036 after multiple doses of ACT-453859 | 11 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. λZ will be determined by log-linear regression analysis of the measured plasma concentrations of the terminal elimination phase.
t1/2 for multiple doses of ACT-453859 | 11 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. t1/2 will be calculated as follows: t½ = ln 2/λZ.
t1/2 for the active metabolite ACT-463036 after multiple doses of ACT-453859 | 11 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. t1/2 will be calculated as follows: t½ = ln 2/λZ.
CLR following multiple doses of ACT-453859 100 mg per day | 8 days
  Urine samples for pharmacokinetic assessments will be collected at various time points over the study period. CLR will be calculated by dividing the total amount of unchanged ACT-453859 excreted in urine during the collection interval by AUC(0-t).
Percentage of ACT-453859 excreted unchanged in the urine following multiple doses of ACT-453859 100 mg per day | 8 days
  Urine samples for pharmacokinetic assessments will be collected at various time points over the study period. The percentage of total dose excreted unchanged in urine will be calculated by the total amount excreted, divided by the dose administered, multiplied by 100.
AUCτ for setipiprant after multiple doses of 500 and 1000 mg b.i.d. setipiprant (Day 1 & Day 7) | 10 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. AUCτ will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the LOQ during one dosing interval.
Cmax for setipiprant after multiple doses of 500 and 1000 mg b.i.d. setipiprant (Day 1 & Day 7) | 10 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. The measured individual plasma concentrations of setipiprant will be used to directly obtain Cmax.
tmax for setipiprant after multiple doses of 500 and 1000 mg b.i.d. setipiprant (Day 1 & Day 7) | 10 days
  Blood samples for pharmacokinetic assessments will be collected at various time points over the study period. The measured individual plasma concentrations of setipiprant will be used to directly obtain tmax.
Chemoattractant receptor-homologous molecule expressed on T helper 2 cells (CRTH2) antagonist pharmacodynamic (PD) effect after single doses of ACT-453859 | 72 hours
  Blood samples for PD assessment will be collected at various time points over the study period. The CRTH2 receptor level on eosinophils and basophils will be measured with flow cytometry and the percentage of eosinophil and basophil CRTH receptors blocked determined.
CRTH2 antagonist PD effect after multiple doses of ACT-453859 | 10 days
  Blood samples for PD assessment will be collected at various time points over the study period. The CRTH2 receptor level on eosinophils and basophils will be measured with flow cytometry and the percentage of eosinophil and basophil CRTH receptors blocked determined.
CRTH2 antagonist PD effect after multiple doses of setipiprant | 10 days
  Blood samples for PD assessment will be collected at various time points over the study period. The CRTH2 receptor level on eosinophils and basophils will be measured with flow cytometry and the percentage of eosinophil and basophil CRTH receptors blocked determined.
CRTH2 antagonist potency following administration of single and multiple doses of ACT-453859 and setipiprant | up to 10 days
  Study drug concentration that elicits 50% blockade (IC50) of eosinophil and basophil CRTH receptors.
Change from baseline up to end of study in systolic blood pressure | up to 11 days
  Blood pressure and heart rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements will be recorded from the subject in the supine and standing position after having rested for a 5-minute period, except for Part C in which only supine position measurements will be performed. Standing position measurements will be performed after one minute standing.
Change from baseline up to end of study in diastolic blood pressure | up to 11 days
  Blood pressure and heart rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements will be recorded from the subject in the supine and standing position after having rested for a 5-minute period, except for Part C in which only supine position measurements will be performed. Standing position measurements will be performed after one minute standing.
Change from baseline up to end of study in heart rate | up to 11 days
  Blood pressure and heart rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements will be recorded from the subject in the supine and standing position after having rested for a 5-minute period, except for Part C in which only supine position measurements will be performed. Standing position measurements will be performed after one minute standing.
Change from baseline up to end of study in QT interval (Time interval from beginning of the Q wave until end of the T wave) | up to 11 days
  Standard 12-lead electrocardiograms will be recorded at rest with the subject in the supine position for at least a 5-minute period at various time points throughout the study.
Change from baseline up to end of study in QTcB interval (QT interval corrected for heart rate according to Bazett's correction) | up to 11 days
  Standard 12-lead electrocardiograms will be recorded at rest with the subject in the supine position for at least a 5-minute period at various time points throughout the study. The QTcB interval is the QT interval corrected for heart rate with Bazett's formula (QTcB = QT/RR^0.5 where RR is 60/heart rate).
Change from baseline up to end of study in QTcF interval (QT interval corrected for heart rate according to Fridericia's correction) | up to 11 days
  Standard 12-lead electrocardiograms will be recorded at rest with the subject in the supine position for at least a 5-minute period at various time points throughout the study. The QTcF interval is the QT interval corrected for heart rate with Fridericia's formula (QTcF = QT/RR^0.33 where RR is 60/heart rate).
Change from baseline up to end of study in heart rate | up to 11 days
  Standard 12-lead electrocardiograms will be recorded at rest with the subject in the supine position for at least a 5-minute period at various time points throughout the study.
Number of subjects with treatment-emergent electrocardiogram abnormalities | up to 11 days
  Standard 12-lead electrocardiograms will be recorded at rest with the subject in the supine position for at least a 5-minute period at various time points throughout the study. Treatment-emergent electrocardiogram abnormalities are defined as abnormalities occurring after study drug administration up to end of study and which were not observed either at pre-dose or screening.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Géhin, PhD, Study Director — Actelion